CLINICAL TRIAL: NCT03954886
Title: Effects of Defocus on Choroidal Thickness
Brief Title: Defocus Induced Changes on Choroidal Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Lisa Ostrin, Assistant Professor, University of Houston
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000852
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Induced Defocus to the Retina
Keywords: Myopia; Choroid; Retina; Blur; Defocus; Eye growth
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Induced myopic defocus (Experimental): Subjects will view a television through a lens that induces blur to the retina for one hour. Images of the eye will be captured every 10 minutes
  Interventions: Device: Plus powered optical lens
- No defocus (No Intervention): Subjects will view a television through a lens that induces no blur to the retina for one hour. Images of the eye will be captured every 10 minutes

INTERVENTIONS:
Device: Plus powered optical lens — A plus powered optical lens will be placed in front of one eye.
  Arms: Induced myopic defocus

SUMMARY:
The goals of this study are to assess the short-term (10-60 minutes) effects of different magnitudes of myopic and hyperopic optical defocus on the transient thickness of the choroid in children and adults, as well as to assess the recovery period. Choroidal thickness will be measured non-invasively following 10-60 minutes of monocular exposure to -5 diopters to +5 diopters of optical defocus induced by spectacle lenses. The hypothesis is that choroidal thickness will increase with increasing myopic defocus and decrease with increasing hyperopic defocus. The relationship between the magnitude of defocus and the magnitude and direction of choroidal thickness change will be assessed.

DETAILED DESCRIPTION:
The purpose of this study is to determine modifying factors inducing or protecting against the development or progression of myopia, or nearsightedness. Myopia has reached epidemic levels in urbanized countries, reaching up to 90% of the teenage and young adult population in urban Asia. Myopia represents a significant socioeconomic burden and poses a risk for associated ocular diseases such as retinal detachment, choroidal neovascularization, and glaucoma. The economic and public health burden of myopia are growing disproportionately to the population, spurring interest in the development of therapies to prevent occurrence or progression. Myopia generally occurs because the eye grows too long, with onset and progression occurring from about ages 6 to 20. Though much is known about factors that influence eye growth, the exact mechanisms by which they do so have not been elucidated.

The goals of this study are to assess the short-term (10-50 minutes) effects of different magnitudes of myopic and hyperopic optical defocus on the transient thickness of the choroid in children and adults, as well as to assess the recovery period. Choroidal thickness will be measured non-invasively following 10-50 minutes of monocular exposure to -5D to +5D of optical defocus induced by spectacle lenses. The hypothesis is that choroidal thickness will increase with increasing myopic defocus and decrease with increasing hyperopic defocus. The relationship between the magnitude of defocus and the magnitude and direction of choroidal thickness change will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 45 years of age (preliminary studies indicate that children under 6 cannot sit for imaging, and subjects over 45 do not respond to the optical defocus with expected choroidal thickness changes)
* Best corrected visual acuity of 20/25 or better in better-seeing eye

Exclusion Criteria:

* Age younger than 6 years or older than 45
* Best corrected visual acuity worse than 20/25 in better-seeing eye
* Ocular pathology or prior ocular injury
* Heavily-pigmented choroid that precludes accurate measurement of choroidal thickness

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | 1 hour
  Changes in choroidal thickness following induced myopic defocus

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be provided by request once published
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At any point after completion of the study and publication